CLINICAL TRIAL: NCT07230340
Title: A Multicenter, Randomized Trial Evaluating Dehydrated Human Placenta Tissue (dHPT) and Standard of Care Versus Standard of Care Alone in Nonhealing Venous Leg Ulcers With Crossover for Subjects Randomized to Standard of Care
Brief Title: Nonhealing Venous Leg Ulcers Treated With a Standard of Care (SoC) Alone or Standard of Care and Dehydrated Human Placenta Tissue (dHPT) With Crossover
Acronym: EVOLVE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cellution Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CELLBIO-2025-002
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Venous Leg Ulcer (VLU)
Keywords: VLU; Venous Ulcer; Leg Wound; Venous Leg Ulcers (VLUs); Amniotic; Placenta; allograft
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Beginning at the screening visit, participants will receive weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 10 weeks, whichever occurs first.
  Interventions: Procedure: Standard of Care (SOC)
- AIC and Standard of Care (Experimental): Participants with a venous leg ulcer (VLU) will receive treatment with an Amnion-Intermediate-Chorion (AIC) sheet product, a dehydrated multilayer human placental tissue derived from donated human tissue, and weekly treatment with standard of care (cleaning, debridement, ulcer moisture balance, and offloading) until ulcer closure, or a maximum of 10 weeks, whichever occurs first.
  Interventions: Other: Amnion-Intermediate-Chorion; Procedure: Standard of Care (SOC)

INTERVENTIONS:
Other: Amnion-Intermediate-Chorion — Dehydrated human placental multilayer allograft derived from donated human tissue. AIC contains amnion and chorion layers as well as basement membrane and trophoblast.
  Arms: AIC and Standard of Care
Procedure: Standard of Care (SOC) — Standard of care is to establish a clean, healthy wound bed and optimize the wound environment to have the best chance of healing the wound. This is achieved through wound cleansing, debridement, offloading and moisture balance.

SUMMARY:
The purpose of this study is to determine how well our dHPT (Dehydrated Human Placental Tissue) Product and Standard of Care work when compared to Standard of Care alone in achieving complete closure of venous leg ulcers.

DETAILED DESCRIPTION:
In 2020, more than 4.5 billion people around the world were estimated to have chronic venous disease stages C1-C6, and approximately 3 in every 1000 people globally develop a VLU annually. While the pathophysiology of VLUs is complex, risk factors are thought to include noncompliance with compression therapy, incorrect ulcer diagnosis, obesity, and a history of deep vein thrombosis. It is estimated that 7% of VLUs do not heal within a 12-month period. As with DFUs, treatment of VLUs focuses on prevention. Low-income individuals, especially those from minority communities, often face difficulties in accessing advanced wound care centers. The estimated annual cost of treating VLUs in the United States in 2022 was over $4.9 billion, which includes expenses for practitioners, wound care products, hospital stays, medications, and compression therapy.

Despite the well-established standard of care for chronic wounds, which includes sharp debridement, offloading, compression therapy, and maintaining proper moisture balance, a notable gap remains between clinical outcomes and desired results in chronic wound care. The reported recurrence rate for venous leg ulcers (VLUs) also ranges from 24% - 57%, illustrating the long-term burden this pathology places on patients.

One approach to treating chronic wounds involves the use of cellular, acellular, and matrix-like products (CAMPs), which are defined as 'A broad category of biomaterials, synthetic materials, or biosynthetic matrices that support repair or regeneration of injured tissues through various mechanisms of action. The application of CAMPs in chronic wound treatment provides several benefits, including creating a protective environment for healing, covering deep structures, aiding surgical closure, enhancing functional outcomes, and improving appearance. The cellular category of CAMPS includes allografts, which are human donor tissue samples intended for use in other human patients. Utilizing dehydrated human placental tissue (dHPT) as an allograft displays considerable promise for chronic wound treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants are required to meet all the following criteria for enrollment into the study:

1. 18 years of age or older.
2. Hemoglobin A1c (HbA1c) level is <12% (108 mmol/mol).
3. Target ulcer with a surface area of between 1.0 cm 2 and 25.0 cm 2 measured post debridement at randomization.
4. Target ulcer must have been present for a minimum of 4 weeks with standard of care prior to the initial screening visit.
5. Affected limb must have adequate perfusion confirmed by vascular assessment performed within 90 days of screening visit. Any of the following methods are acceptable:

   1. ABI ≥ 0.7 and ≤ 1.3;
   2. TBI ≥ 0.6;
   3. TCOM ≥ 40 mmHg;
   4. PVR: biphasic or triphasic.
6. If the participant has two or more ulcers, they must be separated by at least 2 cm post debridement. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.
7. The participant must agree to attend the weekly study visits required by the protocol.
8. The participant must be willing and able to participate in the informed consent process

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from enrollment:

1. Known life expectancy of <6 months.
2. Target ulcer is infected or there is cellulitis in the surrounding skin.
3. Evidence of osteomyelitis complicating the target ulcer.
4. Participant requires systemic antibiotic therapy or has used within the last 7 days.
5. Receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent), receiving cytotoxic chemotherapy, or taking medications that the investigator believes will interfere with wound healing (e.g., biologics).
6. Topical application of steroids to the ulcer surface within 30 days of screening.
7. Target ulcer exposes tendon or bone.
8. Surface area of the target ulcer decreases by more than 20% during the 2-week screening phase.
9. Mini Nutritional Assessment (MNA) score of less than 17.
10. Participants of child bearing potential who are pregnant, considering becoming pregnant within the next 6 months, and/or are unwilling to utilize an appropriate form of contraception.
11. Currently requiring dialysis or planning to start within 6 months.
12. Medical or psychological condition that, in the opinion of the investigator, may interfere with study assessments.
13. Treated with hyperbaric oxygen therapy or a skin substitute within the 30 days prior to screening visit.
14. Sensitivity to ofloxacin, vancomycin, or amphotericin antibiotics.
15. Participation in a clinical trial involving treatment with an investigational product within the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Venous Leg Ulcers with Complete Wound Closure | 1-10 weeks
  The percentage of VLU target ulcers achieving complete wound closure. Closure is defined as 100% re-epithelialization of the ulcer surface without detectable exudate.

SECONDARY OUTCOMES:
Time to Complete Closure for Ulcer | 1-10 weeks
  Time to closure will be determined for the treatment group and compared to Standard of Care. Closure is defined by 100% re-epithelialization of the ulcer surface without detectable exudate.
Percentage of Wound Area Change for Target Ulcer | 1-10 weeks
  Percentage wound area changes from week 1 to week 10 will be calculated weekly from measurements with digital photographic images and physical examination.
Incidents of Adverse Events | 1-10 weeks
  Changes in quality of life using both the Wound Quality of Life (wQOL) and Forgotten Wound Score (FWS) questionnaires that measure the health-related quality of life (HRQoL) of patients with chronic wounds. wQOL questionnaire is scored using a 5-point Likert scale, where 0 means "not at all" and 4 means "very much". Higher scores indicate greater impairment of quality of life. Higher the score indicates lower quality of life. FWS questionnaire measures 12 activities scored 0-4. Responses are summed and divided by the number of completed items. The mean value is then multiplied by 25 to obtain the total score of 0-100. Higher the score indicates lower quality of life.

OTHER OUTCOMES:
Changes in Pain Associated with the Target Ulcer | 1-10 weeks
  Change in pain in the target ulcer assessed using the Visual Analog Scale (VAS) from week 1 to week 10. VAS is a tool that uses a 0-10 (no o extreme pain) point scale to measure pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Research Director, Study Director — Cellution Biologics

IPD SHARING:
Plan to Share IPD: No